CLINICAL TRIAL: NCT03883191
Title: Effect of a Three Combined Probiotics Supplementation on Weight Loss in Obese/Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, An-Chyi Chen, Principal Investigator, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH105-REC2-096
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Obesity, Childhood
Keywords: Probiotics; Overweight; Obese; Children; Weight reduction
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Probiotic or placebo group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mix probiotics powder (Experimental): Taking 1 pack of L. rhamnosus bv-77, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics powder three times a day before meals for three months.
  Interventions: Other: L. rhamnosus bv-77, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics powder
- Placebo powder (Placebo Comparator): Taking 1 pack of placebo powder three times a day before meals for three months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: L. rhamnosus bv-77, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics powder — Taking 1 pack of L. rhamnosus bv-77, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics powder three times a day before meals for three months.
  Arms: Mix probiotics powder
Other: Placebo — Taking 1 pack of placebo powder three times a day before meals for three months.
  Arms: Placebo powder

SUMMARY:
This program is a double-blind, randomized, placebo-controlled study. Investigators expect to enroll 100 overweight or obese children those ages 6 to 18 years. A product that containing three probiotics will be prescribed for study group for 12 weeks plus diet and exercise guidance, while the control group will be given a placebo plus diet and exercise guidance.

DETAILED DESCRIPTION:
The prevalence of obesity in adults was up to 40% in Taiwan. The prevalence of overweight and obesity in Taiwanese boy was over 30%, while close to 30% of Taiwanese girls were overweight and obesity. Obese children are more prone to becoming obese adults and consequently increased risk of many complications, including metabolic syndrome, nonalcoholic fatty liver disease, cardiovascular disease, etc. Therefore, childhood obesity may result in significant public health burden in the future if it was improperly handled. Unfortunately, there is still lack of effective way to reduce weight and long-term weight control except for lifestyle modification.

Recent studies have shown that microflora of the gut are associated with obesity, perhaps one of the cause of obesity. Many studies have shown that the gut microbiota is different between obese individuals and normal-weight individuals. The most significant one is that obese individuals have larger Firmicutes/Bacteroidetes ratio. In the other hand, many studies have confirmed that probiotic was effectively in weight loss in obese adults. However, there are only few research in pediatric population in this issue. Researchers have demonstrated that products containing probiotics are effective in reducing weight, BMI, and serum lipid level in obese child.

This program is a double-blind, randomized, placebo-controlled study. Investigators expect to enroll 100 overweight or obese children those ages 6 to 18 years. A product that containing three probiotics will be prescribed for study group for 12 weeks plus diet and exercise guidance, while the control group will be given a placebo plus diet and exercise guidance. Every subjects will receive several tests and examinations before and after the study, such as: height, weight, BMI, waist circumference, body fat, blood pressure, blood sugar, blood lipids profile, liver and kidney function, and abdominal ultrasound. Investigators will compare these parameters between these two groups after the study. Investigators expect to follow these subjects for more than one year, to see if this product has persistent effects.

ELIGIBILITY:
Inclusion Criteria:

1. Over 6 years old under 18 years old.
2. Overweight or obese children without potential disease.Overweight or obese children is defined by the "Children's and Adolescent Growth Body Mass Index (BMI) Recommended Values" published by the National Health Agency of the Ministry of Health and Welfare on June 11, 2013.

Exclusion Criteria:

1. There are major potential diseases, such as congenital heart disease, severe asthma, chronic hepatitis, renal dysfunction, neurodegenerative diseases and major genetic diseases.
2. Drugs such as weight loss drugs, hypolipidemic drugs, hypoglycemic agents, blood pressure lowering drugs, oral steroids, and hormone supplements are being used.
3. Those who use probiotics or related products for a long time.
4. Those who use antibiotics during the test.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Change in the body mass index (BMI) after intervention | Up to 3 months.
  Body weight (kg) and height (m) will be combined to report BMI in kg/m^2, normal BMI value is defined by the "Children's and Adolescent Growth Body Mass Index Recommended Values" published by the National Health Agency of the Ministry of Health and Welfare on June 11, 2013. Probiotics and placebo group BMI value will be presented as an average, lower values represent a better outcome.
Change in the waist circumference after intervention | Up to 3 months.
  Waist circumference in centimeters, probiotics and placebo group waist circumference value will be presented as an average, lower values represent a better outcome.
Change in the body fat after intervention | Up to 3 months.
  Body fat (%) in percentage of body weight, probiotics and placebo group body fat percentage will be presented as an average, lower values represent a better outcome.
Change in the blood pressure after intervention | Up to 3 months.
  Blood pressure in mmHg, probiotics and placebo group blood pressure value will be presented as an average, lower values represent a better outcome.
Change in the blood sugar and blood lipids after intervention | Up to 3 months.
  Blood sugar and blood lipids in mg/dl, probiotics and placebo group blood sugar and blood lipids value will be presented as an average, lower values represent a better outcome.
Change in the liver function after intervention | Up to 3 months.
  Liver function is defined as glutamic oxaloacetic transaminase (GOT) and glutamic pyruvic transaminase (GPT) in IU/L, probiotics and placebo group GOT and GPT value will be presented as an average, lower values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-chih Lin, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan